CLINICAL TRIAL: NCT04320199
Title: Effect of Fermented Protaetia Brevitarsis Seulensis Powder on Alcohol-induced Liver Disease: a Randomized Controlled Trial
Brief Title: Effect of Fermented Protaetia Brevitarsis Seulensis Powder on Alcohol-induced Liver Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2018-025
Record Dates: First submitted 2020-03-21; First posted 2020-03-24 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Alcoholic Liver Disease
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fermented Protaetia brevitarsis seulensis powder group (Experimental): This group takes Fermented Protaetia brevitarsis seulensis powder for 8 weeks
  Interventions: Dietary Supplement: Fermented Protaetia brevitarsis seulensis powder group
- Placebo group (Placebo Comparator): This group takes placebo for 8 weeks
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Fermented Protaetia brevitarsis seulensis powder group — This group takes Fermented Protaetia brevitarsis seulensis powder for 8 weeks
  Arms: Fermented Protaetia brevitarsis seulensis powder group
Dietary Supplement: Placebo group — This group takes placebo for 8 weeks
  Arms: Placebo group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Fermented Protaetia brevitarsis seulensis powder on Alcohol-induced Liver Disease in adults for 8 weeks.

DETAILED DESCRIPTION:
Previous studies have indicated that Fermented Protaetia brevitarsis seulensis powder may have the ability to improve liver function in adults with alcohol-induced liver disease. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Fermented Protaetia brevitarsis seulensis powder on liver function in adults with alcohol-induced liver disease; the safety of the compound are also evaluate. The Investigators examine gamma-glutamyl transferase, alanine aminotransferase, aspartate aminotransferase, and other metabolic parameters at baseline, as well as after 4 and 8 weeks of intervention. Sixty adults were administered either 4,000 mg of Fermented Protaetia brevitarsis seulensis powder or a placebo each day for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Gamma-glutamyl transferase ranging from upper limit of reference to four times of upper limit

Exclusion Criteria:

* Abnormal liver or renal function (i.e., serum aminotransferase activity > 3 times of upper limit of reference range and serum creatinine concentrations > 1.2 mg/dL)
* Diabetes (diagnosed clinically or fasting glucose level > 126 mg/dL)
* History of viral hepatitis or cancer
* Uncontrolled hypertension
* History of serious cardiac disease such as angina or myocardial infarction
* History of gastrectomy
* History of medication for psychiatric disease
* Administration of oriental medicine including herbs within the past 4 weeks

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of Gamma-Glutamyl Transpeptidase | 8 weeks
  Gamma-Glutamyl Transpeptidase

SECONDARY OUTCOMES:
Concentration of Aspartate aminotransferase | 8 weeks
  Aspartate aminotransferase
Concentration of Alanine aminotransferase | 8 weeks
  Alanine aminotransferase
Fatigue Severity Scale | 8 weeks
  Fatigue Severity Scale, minimum~maximum values (1~7), higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, Professor, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Pusan, Ami-dong, South Korea

IPD SHARING:
Plan to Share IPD: No